CLINICAL TRIAL: NCT00342160
Title: Virologic and Immunologic Factors Contributing to the Lack of HIV-1 Transmission in HIV-Discordant Couples in Rakai, Uganda
Brief Title: Viral and Immunologic Factors Contributing to the Lack of HIV Transmission Among Couples in Rakai, Uganda
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906100; 06-I-N100
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-11-13

CONDITIONS: HIV
Keywords: AIDS; HIV Infectiousness; Immunity; CTL; Epidemiology
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

SUMMARY:
This study will look at viral and immunologic factors involved in protecting against sexually transmitted HIV infection in couples in which one partner is infected and the other is not.

This study will include 50 couples who reside in Rakai, Uganda, and who have been together for at least 2 years. In some couples, both partners will be HIV-infected, in some couples only one partner will have HIV, and in some couples neither partner will have HIV.

Participants undergo the following procedures at each of four study visits:

* HIV counseling and testing
* Medical history, including questions about personal behaviors such as sexual practices and use of condoms
* Blood sample collection
* Urine sample collection
* Vaginal swab for women

Blood, urine and vaginal fluid samples are tested for HIV and other sexually transmitted diseases, such as syphilis. Blood and vaginal samples are also tested for HIV viral levels and immune response in HIV-infected individuals and for evidence of exposure to HIV in non-infected participants. Some blood is also tested for genetic markers to investigate whether certain proteins are related to resistance to HIV infection.

...

DETAILED DESCRIPTION:
Understanding the factors that contribute to the transmission of human immunodeficiency virus (HIV) infection is of great importance for the development of preventive and therapeutic strategies. Evidence suggests that a number of host immunologic and virologic factors play critical roles in protection against sexually transmitted HIV infection in HIV-discordant partners. Among these, the antiviral role of CD8+ T cells in HIV-infected individuals has been extensively studied. At least two types of CD8+ T cell-mediated antiviral activities have been described in HIV infection. The first is a suppressive activity against HIV involving lysis of infected cells in an antigen-specific, HLA-restricted fashion, while the second mechanism inhibits viral replication via either cell- or soluble mediated factors in the absence of cell killing. It has been demonstrated that cytotoxic CD8+ T lymphocytes (CTL) are present in both cervical and peripheral blood mononuclear cells (PBMC) from a subpopulation of highly-HIV-exposed but persistently seronegative individuals. However, studies addressing the effect of non-cytotoxic soluble factor-mediated antiviral activity by CD8+ T cells in preventing seroconversion in HIV-discordant couples have been lacking. This study proposes to examine the role of CD8+ T cell-derived CC-chemokine activities and the copy numbers of one of the chemokine genes, CCL3L1, along with other host anti-HIV and virologic factors in resistance to HIV infection in persistently seronegative HIV-discordant partners of HIV infected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group 1 (HIV concordant partners, n = 20 couples):

* Documentation of HIV infection in both partners, a current history of continued sexual activity within the partnership, and demonstration that they have been in a partnership for at least two years.
* CD4+ T cell count greater than 250/microliters blood in both partners and not currently on HAART.
* Plasma viremia greater than 5,000 copies of HIV RNA/ml plasma in both partners.
* Able and willing to provide informed consent.
* Must agree to continued couple counseling regarding HIV results

Group 2 (HIV-discordant partners, n = 20 couples):

* Documentation of HIV infection in one partner and seronegative status in the other partner, a current history of continued sexual activity within the partnership, and demonstration that they have been in a partnership for at least two years.
* CD4+ T cell count greater than 250/microliters blood in both partners and not currently on HAART.
* Plasma viremia greater than 5,000 copies of HIV RNA/ml plasma in each infected partner.
* Able and willing to provide informed consent.
* Must agree to continued couple counseling regarding HIV results

Group 3 (HIV-uninfected partners, n = 10 couples):

* Documentation of HIV-seronegative status in both partners, a current history of continued sexual activity within the partnership, and demonstration that they have been in a partnership for at least two years.
* CD4+ T cell count greater than 250/microliters blood in both partners.
* Able and willing to provide informed consent.
* Must agree to continued couple counseling regarding HIV results

EXCLUSION CRITERIA:

Inability or unwillingness to provide individual informed consent, on the part of either or both members of the couple.

Refusal of couples counseling on the part of one or both partners.

Severe illness in one or the other, and /or a hemoglobin value less than 8 g/dL.

Age less than 18. Children are not included in this study since it specifically focuses on sexual transmission of HIV in long term married couples.

Having had a blood transfusion within the last 60 days. Though individuals can be scheduled after this time period has passed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-02-15; Study Completion 2012-11-13

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Quinn, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Uganda Virus Research Institute, Rakai, Uganda

REFERENCES:
- [Background] Blocker ME, Cohen MS. Biologic approaches to the prevention of sexual transmission of human immunodeficiency virus. Infect Dis Clin North Am. 2000 Dec;14(4):983-99. doi: 10.1016/s0891-5520(05)70143-4. PMID 11144648
- [Background] Quinn TC, Wawer MJ, Sewankambo N, Serwadda D, Li C, Wabwire-Mangen F, Meehan MO, Lutalo T, Gray RH. Viral load and heterosexual transmission of human immunodeficiency virus type 1. Rakai Project Study Group. N Engl J Med. 2000 Mar 30;342(13):921-9. doi: 10.1056/NEJM200003303421303. PMID 10738050
- [Background] Vernazza PL, Troiani L, Flepp MJ, Cone RW, Schock J, Roth F, Boggian K, Cohen MS, Fiscus SA, Eron JJ. Potent antiretroviral treatment of HIV-infection results in suppression of the seminal shedding of HIV. The Swiss HIV Cohort Study. AIDS. 2000 Jan 28;14(2):117-21. doi: 10.1097/00002030-200001280-00006. PMID 10708281